CLINICAL TRIAL: NCT06094634
Title: IGHID 12219 - A Brief Alcohol Intervention to Reduce Alcohol Use and Improve PrEP Outcomes: A Randomized Controlled Trial
Brief Title: IGHID 12219 - A Brief Alcohol Intervention for PrEP Users
Acronym: BPrEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institutes of Health (NIH) (NIH); Hanoi Medical University (Other); Johns Hopkins University (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23-0256; R01AA030479 (NIH)
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Unhealthy Alcohol Use
Keywords: Preexposure Prophylaxis (PrEP); Alcohol Intervention; Motivational Interviewing; Cognitive Behavioral Therapy; Motivational Enhancement Therapy; Cost Analysis; Economic Evaluation
MeSH Terms: interventions — Ethanol; Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assessment-only control (No Intervention): Participants receive study assessment visits and standard of care from providers at the PrEP clinic.
- The Brief Alcohol Intervention (BAI) (Experimental): Participants receive the Brief Alcohol Intervention (2 in-person sessions and 2 phone sessions), study assessment visits, and standard of care from providers at the PrEP clinic.
  Interventions: Behavioral: The Brief Alcohol Intervention (BAI): Behavioral

INTERVENTIONS:
Behavioral: The Brief Alcohol Intervention (BAI): Behavioral — The BAI draws from Motivational Interviewing (MI)/Motivational Enhancement Therapy (MET) and Cognitive Behavioral Therapy (CBT) and comprises 2 in-person face-to-face sessions and 2 booster telephone sessions by a trained counselor.
  Arms: The Brief Alcohol Intervention (BAI)

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a brief alcohol intervention (BAI) vs. standard of care (SOC) to improve pre-exposure prophylaxis (PrEP) use among PrEP initiators and re-initiators.

DETAILED DESCRIPTION:
This is a two-arm effectiveness randomized controlled trial (RCT) to compare the brief alcohol intervention (BAI) to the standard of care (SOC) among PrEP initiators and re-initiators with unhealthy alcohol use who are initiating or reinitiating oral, event-driven, or injectable PrEP.

The BAI draws from Motivational Interviewing (MI)/Motivational Enhancement Therapy (MET) and Cognitive Behavioral Therapy (CBT) and includes 2 in-person sessions and 2 telephone sessions.

Eligible participants (n=564) will be randomized 1:1 to each arm (282 per arm). Additional assessments among a subset of participants in the BAI arm will assess acceptability of the intervention (n=48).

Study activities will span 5 years. Individual PrEP initiators and re-initiators will be followed-up for 12 months with assessment visits at 3, 6, 9, and 12 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Newly initiating PrEP or re-initiating PrEP after at least 3 months from a missed PrEP appointment, based on local PrEP guidelines
* AUDIT-C score ≥ 4 or CRAFFT score ≥ 2 (for those ≤21 years old)
* 16 years of age or older
* Intention to receive PrEP care in Hanoi for 12 months
* Willingness to provide informed consent

Exclusion Criteria:

* Psychological disturbance, cognitive impairment, or threatening behavior
* Unwilling to provide locator information
* Current participation in alcohol programs or studies
* Current participation in other research studies (including HIV and PrEP studies)
* Ever enrolled in an HIV vaccine study
* Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA) ≥ 10, indicating risk for alcohol withdrawal

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
PrEP Persistence | 12 months
  PrEP persistence is a measure of ongoing PrEP usage, defined as consistent presentation for care and refills.
Heavy Drinking Days (Binge drinking) | 12 months
  The number of days with ≥6 standard drinks of alcohol per occasion among the previous 30 days as assessed on the Timeline Followback.
Incremental Cost-Effectiveness Ratio (ICER) | 12 months
  The incremental cost-effectiveness ratio (ICER) is expressed as the incremental cost of the Brief Alcohol Intervention (BAI) per quality adjusted life-year (QALY) gained. ICER is defined as [Ci - Ca]/[Ei - Ea] with Ci and Ca being the respective costs of the BAI [i] and assessment only [a], and Ei and Ea the corresponding effectiveness.
Acceptability of the brief alcohol intervention, as measured with mHIST | 3 months
  Acceptability is an implementation-focused outcome and will be assessed using the Mental Health Implementation Science Tools (mhIST) Acceptability Scale for consumers, which consists of 15 items containing responses on a 4-point Likert scale. The mhIST score is calculated as the mean score of all responses ranging from 0-3. Higher mhIST scores indicate higher acceptability.
Feasibility - proportion completed 4 sessions (intervention arm) | 17 weeks
  Feasibility is an implementation-focused outcome and will be measured as the BAI completion rate among participants. Three metrics will be considered. The first metric will be the proportion of participants who completed all 4 sessions among those who were assigned to the intervention arm, measured from the date of randomization.
Feasibility - proportion completed 2 sessions (intervention arm) | 17 weeks
  Feasibility is an implementation-focused outcome and will be measured as the BAI completion rate among participants. Three metrics will be considered. The second metric will be the proportion of participants who completed at least 2 sessions among those who were assigned to the intervention arm, measured from the date of randomization.
Feasibility - proportion completed 4 sessions (among initiators) | 10 weeks
  Feasibility is an implementation-focused outcome and will be measured as the BAI completion rate among participants. Three metrics will be considered. The third metric will be the proportion of participants who completed at least 4 sessions among those who initiated at least one session, measured from the date of the first in-person session.

SECONDARY OUTCOMES:
PrEP Adherence | Up to 12 months
  PrEP adherence is a measure of pill-taking behavior and will be assessed by self-report and pharmacy records. Adherence will be assessed per person based on the type of PrEP prescribed but will be compared as a single measure.
  Oral and event-driven PrEP adherence will be assessed as self-reported number of doses taken.
  Oral PrEP adherence is defined with two thresholds: ≥ 4 days/week, a threshold consistent with standard prevention definitions, and 7 days/week, indicating perfect adherence.
  Event-driven PrEP adherence will be defined as completion of the 2+1+1 regimen for every reported intercourse event.
Risk-aligned PrEP use | Up to 12 months
  Risk-aligned PrEP use is a measure of whether PrEP use is consistent with concurrent risk behavior. It is defined as persistent oral/injectable PrEP, event-driven PrEP (2+1+1), or clinician-supervised PrEP discontinuation.
  More specifically, risk-aligned PrEP is defined as:
  1. Persistent oral, event-driven or injectable PrEP,
  2. Clinician-approved PrEP discontinuation.
Number of Drinking Days | Up to 12 months
  Number of drinking days is defined as the number of days with any alcohol use, among the previous 30 days as assessed on the Timeline Followback. The timeline followback will be administered at enrollment, 3 months and 12 months.
Number of Drinks Per Drinking Day | Up to 12 months
  Drinks per drinking day is defined as the number of standard drinks of alcohol consumed on a drinking day, among the past 30 days as assessed on the Timeline Followback. The timeline followback will be administered at enrollment, 3 months and 12 months.
Penetration | Up to 7 weeks
  Completion of at least one session among those assigned to the intervention arm, measured from the date of randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian F Go, PhD, Principal Investigator — University of North Carolina; William C Miller, MD, PhD, Principal Investigator — University of North Carolina; Le Minh Giang, MD, PhD, Principal Investigator — Hanoi Medical University
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Bui HTM, Giang LM, Chen JS, Sripaipan T, Nong HTT, Nguyen NTK, Bartels SM, Rossi SL, Hutton H, Chander G, Sohn H, Ferguson O, Tran HV, Nguyen MX, Nguyen KD, Rutstein SE, Levintow S, Hoffman IF, Powell BJ, Pence BW, Go VF, Miller WC. A Brief Alcohol Intervention (BAI) to reduce alcohol use and improve PrEP outcomes among men who have sex with men in Vietnam: study protocol for a randomized controlled trial. Trials. 2024 Aug 21;25(1):552. doi: 10.1186/s13063-024-08382-5. PMID 39164770

DOCUMENTS (1):
  • Informed Consent Form (2025-03-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT06094634/ICF_000.pdf